CLINICAL TRIAL: NCT01166555
Title: Phase I Pharmacokinetics And Tolerability Of PF-04236921 Following Subcutaneous Administration To Healthy Volunteers
Brief Title: Pharmacokinetics And Tolerability Of Subcutaneous Administration Of PF 04236921 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: B0151004; EudraCT 2010-019770-32
Record Dates: First submitted 2010-05-11; First posted 2010-07-21 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Safety and tolerability; Pharmacokinetics; PF-04236921; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — PF-04236921

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-04236921

INTERVENTIONS:
Drug: PF-04236921 — single subcutaneous dose

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of PF-04236921 administered as a single subcutaneous dose in healthy volunteers.

DETAILED DESCRIPTION:
Tolerability and Pharmacokinetics of subcutaneously administered dose of PF-04236921 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18-55 years, inclusive.
* Healthy females of non-childbearing potential between 18 and 55 years, inclusive.

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* Females of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 5 months
Incidence and severity of clinical findings on physical examination | 5 months
Mean change from baseline in vital signs (blood pressure, pulse rate, oral or tympanic temperature) measurements | 5 months
Mean change from baseline in 12-lead electrocardiogram (ECG) parameters: PRI, RR, QRS, QT, QTcF (Freidericia's correction) and HR (heart rate) | 5 months
Serum PF-04236921 concentrations will be determined by a validated assay and noncompartmental PK parameters | 5 months

SECONDARY OUTCOMES:
Incidence and severity of clinical laboratory abnormalities including absolute neturophil count, hepatic transaminases and bilirubin levels, and lipid profiles | 5 months
Incidence and level of ADA development | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Li C, Shoji S, Beebe J. Pharmacokinetics and C-reactive protein modelling of anti-interleukin-6 antibody (PF-04236921) in healthy volunteers and patients with autoimmune disease. Br J Clin Pharmacol. 2018 Sep;84(9):2059-2074. doi: 10.1111/bcp.13641. Epub 2018 Jun 25. PMID 29776017
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0151004&StudyName=Pharmacokinetics%20And%20Tolerability%20Of%20Subcutaneous%20Administration%20Of%20PF%2004236921%20In%20Healthy%20Volunteers